CLINICAL TRIAL: NCT06918639
Title: Effectiveness of Pulpotomy in Symptomatic Permanent Teeth With Deep Caries Lesions
Status: Recruiting | Type: Observational
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, OLGA GONZÁLEZ CASTRO, Student of the International Doctoral School, Universidad Rey Juan Carlos, Universidad Rey Juan Carlos
Other Study IDs: 100120240392024
Record Dates: First submitted 2024-06-27; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Irreversible Pulpitis; Pulpotomy of Permanent Molars
Keywords: pulpotomy; vitalpulptherapy; partialpulpotomy; biodentinexp; fullpulpotomy; completepulpotomy
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- to determinate the success of partial and total pulpotomy in permanent teeth: The main outcome of the present study will be the success rate of the treatment, determined by the absence of symptoms of irreversible pulpitis and the absence of radiological images compatible with pathology. The type of pulpotomy (partial or total) to be performed on each tooth will not be randomised for ethical reasons but, unlike other studies, will be determined clinically at the time of treatment according to the indication. Subsequently, the success of each treatment will be compared.
  Interventions: Procedure: Pulpotomy

INTERVENTIONS:
Procedure: Pulpotomy — VPT: Partial pulpotomy: 2 mm of pulp tissue is removed with a high speed 014 diamond round bur different from the one used to remove carious tissue. In those cases in which access to the pulp tissue induces a painful sensation due to failure of the anaesthetic technique, intrapulpal anaesthesia shall be used, and this parameter shall be recorded.Cotton wool impregnated with 2.5% stabilised sodium hypochlorite shall be held over the pulp exposure to achieve haemostasis. If it is not possible to control bleeding, proceed to a complete pulpotomy procedure. If in this case it is impossible to achieve haemostasis, the possibility of performing a TPV is ruled out and the RCT is excluded from the study. Once haemostasis has been achieved, BiodentineXp is applied according to the manufacturer's instructions and a material thickness of 2-3 mm is ensured. Full pulpotomy: The same anterior procedure .Complete removal of the tissue from the pulp chamber. Maximum haemostasis time: 10 minutes

SUMMARY:
Preservation of pulp tissue would allow it to continue to exert its defensive and physiological functions and more tooth tissue would be preserved, leading to less weakening of the tooth. In addition, root canal treatment is a more complex therapeutic process that requires the use of more instruments, more time and more visits. To date, most clinical studies that have evaluated the success of pulpotomy treatments have been conducted on teeth with immature apexes. More studies are needed to evaluate VPT success in the permanent dentition in the long term.

In accordance with the above, the main objective of the study will be to determine the success of partial or total pulpotomy treatment in permanent teeth (>18 adults) with a closed apex and symptoms compatible with irreversible pulpitis. At the same time, the association of factors related to the patient, the treated tooth and specific treatment factors with the success of pulpotomies will be determined. On the other hand, the patient, perception and satisfaction with the treatment received will be evaluated.

All treatments (pulpotomies and restorations) will be carried out by the principal investigator.

After recording the preoperative data, clinical and radiographic examination, a diagnosis will be made according to the classification of Wolters and collaborators , which will also guide us in the choice of pulp treatment: PP o CP Partial pulpotomy or complete pulpotomy. The maximum pulp haemostasis time will be 10 minutes. In both treatments, in the same appointment, the definitive restoration of the tooth will be carried out.

The evaluations will be performed at one week, 3 , 6 and 12 months postoperatively. This evaluation shall be performed by an examiner who shall be different from the one performing the treatment.

The main outcome of the present study will be the determination of the success of the pulpotomies.

- Is vital pulp therapy a highly successful treatment for teeth with irreversible pulpitis?.

Outcome measure 1: Success rate of vital pulp therapy

- Do patients feel satisfied with this conservative pulp treatment? Outcome measure 2: Patient´s satisfaction with vital pulp therapy

DETAILED DESCRIPTION:
Success shall be determined by the absence of signs and symptoms in addition to maintenance of pulp vitality. The presence of symptoms compatible with the presence of pulp pathology or the observation of pathological radiolucent lesions will indicate the need for root canal treatment and will be considered failure of vital pulp therapy treatment.

After completion of the procedure, a patient survey will be given to the patient to record the patients, perception and satisfaction with the treatment received.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients in good general health, ASA I or ASA II with no contraindications to contraindications to receive a TPV procedure under local anaesthesia.
* Tooth with symptomatology of pulpitis, both reversible and irreversible, to be determined by history of spontaneous pain, exacerbation of pain with heat and cold confirmed by the cold test and radiating pain.
* Tooth without signs of pulp necrosis and absence of sinus tract and abscess.
* Tooth in occlusion with antagonist tooth and without discomfort on chewing.
* Tooth that can be directly restored.
* Tooth with pocket depth and mobility within normal limits.
* Extent of the caries lesion greater than two thirds of the amelodentine distance or which tooth or the pulp has been exposed during caries removal.

Exclusion Criteria:

* Patients with allergies or intolerance to any anaesthetic solution.
* Pregnant patients or patients who suspect pregnancy due to the impossibility of complementary radiographic tests cannot be carried out.
* Patients with systemic pathology that prevents the use of a vasoconstrictor or with a compromised immune system that may influence the response to treatment.
* Tooth with an immature apex.
* Tooth that is not restorable or not viable for preservation.
* Tooth with negative response to thermal sensitivity test or electrical test.
* Tooth in which haemostasis cannot be achieved after exposure of the pulp, or with a pulp, or with a haemostasis time exceeding 10 minutes, where there is no pulp bleeding or partial or complete tissue necrosis is observed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients (a minimum of 50 teeth, based on previous studies evaluating the success of pulpotomies requiring partial pulpotomy or complete pulpotomy treatment in permanent teeth with closed apex, with symptomatology of pulpitis, both reversible and irreversible, who meet the remaining inclusion criteria, will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of the vital pulpt treatment | From the treatment to the one-year follow-up.
  The evaluation will be according to clinical and radiographic parameters:
  * Clinical: absence of spontaneous pain, normal probing depth, no movility, no sinus tract or swelling.
  * Radiographic findings: No periapical lesions.

SECONDARY OUTCOMES:
Patient satisfaction with vital pulp treatment | From enrollement to the first control visit, 7 days later
  A specific questionnaire has been designed in which patients are asked about the characteristics of the pain before the treatment and 24 hours, 3 and 7 days afterwards, using a visual rating scale. The values ranged between 0 and 10, being 0 the absence of pain and 10 the maximum pain. Moreover, they were also asked regarding the treatment impact on esthetics, function and comfort. Also, a numerical rating scale was used, ranging from 1 to 10, being 10 the maximum satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ceballos, Full Professor, DDS, PhD, Study Director — Universidad Rey Juan Carlos; Victoria Fuentes, Associate Professor, DDS, PhD, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Rey Juan Carlos University, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Careddu R, Plotino G, Cotti E, Duncan HF. The management of deep carious lesions and the exposed pulp amongst members of two European endodontic societies: a questionnaire-based study. Int Endod J. 2021 Mar;54(3):366-376. doi: 10.1111/iej.13418. Epub 2020 Oct 19. PMID 32970860
- [Background] Wolters WJ, Duncan HF, Tomson PL, Karim IE, McKenna G, Dorri M, Stangvaltaite L, van der Sluis LWM. Minimally invasive endodontics: a new diagnostic system for assessing pulpitis and subsequent treatment needs. Int Endod J. 2017 Sep;50(9):825-829. doi: 10.1111/iej.12793. No abstract available. PMID 28776717
- [Background] Ramani A, Sangwan P, Tewari S, Duhan J, Mittal S, Kumar V. Comparative evaluation of complete and partial pulpotomy in mature permanent teeth with symptomatic irreversible pulpitis: A randomized clinical trial. Int Endod J. 2022 May;55(5):430-440. doi: 10.1111/iej.13714. Epub 2022 Mar 10. PMID 35226769
- [Background] Jassal A, Nawal RR, Yadav S, Talwar S, Yadav S, Duncan HF. Outcome of partial and full pulpotomy in cariously exposed mature molars with symptoms indicative of irreversible pulpitis: A randomized controlled trial. Int Endod J. 2023 Mar;56(3):331-344. doi: 10.1111/iej.13872. Epub 2022 Dec 4. PMID 36403208
- [Background] Esteve-Pardo G, Barreiro-Gabeiras P, Esteve-Colomina L. Pulpectomy vs. Pulpotomy as Alternative Emergency Treatments for Symptomatic Irreversible Pulpitis-A Multicenter Comparative Randomised Clinical Trial on Patient Perceptions. Clin Pract. 2023 Aug 2;13(4):898-913. doi: 10.3390/clinpract13040082. PMID 37623263
- [Background] Hickel R, Mesinger S, Opdam N, Loomans B, Frankenberger R, Cadenaro M, Burgess J, Peschke A, Heintze SD, Kuhnisch J. Revised FDI criteria for evaluating direct and indirect dental restorations-recommendations for its clinical use, interpretation, and reporting. Clin Oral Investig. 2023 Jun;27(6):2573-2592. doi: 10.1007/s00784-022-04814-1. Epub 2022 Dec 12. PMID 36504246
- [Background] Taha NA, Abdelkhader SZ. Outcome of full pulpotomy using Biodentine in adult patients with symptoms indicative of irreversible pulpitis. Int Endod J. 2018 Aug;51(8):819-828. doi: 10.1111/iej.12903. Epub 2018 Feb 27. PMID 29397003
- [Background] Taha NA, Al-Khatib H. 4-Year Follow-up of Full Pulpotomy in Symptomatic Mature Permanent Teeth with Carious Pulp Exposure Using a Stainproof Calcium Silicate-based Material. J Endod. 2022 Jan;48(1):87-95. doi: 10.1016/j.joen.2021.09.008. Epub 2021 Sep 24. PMID 34563506
- [Background] Taha NA, Abuzaid AM, Khader YS. A Randomized Controlled Clinical Trial of Pulpotomy versus Root Canal Therapy in Mature Teeth with Irreversible Pulpitis: Outcome, Quality of Life, and Patients' Satisfaction. J Endod. 2023 Jun;49(6):624-631.e2. doi: 10.1016/j.joen.2023.04.001. Epub 2023 Apr 19. PMID 37080387
- [Background] Ricucci D, Siqueira JF Jr, Li Y, Tay FR. Vital pulp therapy: histopathology and histobacteriology-based guidelines to treat teeth with deep caries and pulp exposure. J Dent. 2019 Jul;86:41-52. doi: 10.1016/j.jdent.2019.05.022. Epub 2019 May 21. PMID 31121241
- [Background] Smith AJ, Duncan HF, Diogenes A, Simon S, Cooper PR. Exploiting the Bioactive Properties of the Dentin-Pulp Complex in Regenerative Endodontics. J Endod. 2016 Jan;42(1):47-56. doi: 10.1016/j.joen.2015.10.019. PMID 26699924